CLINICAL TRIAL: NCT03417336
Title: Multicenter, Randomized, Pilot Study Evaluating the Efficacy and the Tolerance of Pelvic-prostatic Hypo-fractionated Radiotherapy Followed by Boost (Stereotaxic External Radiotherapy or High Dose Rate Brachytherapy) in Patients With Prostate Adenocarcinoma Adverse Intermediate Risk or High Localized Risk
Brief Title: Study Evaluating the Efficacy and the Tolerance of Pelvic-prostatic Hypo-fractionated Radiotherapy Followed by Boost in Patients With Prostate Adenocarcinoma Adverse Intermediate Risk or High Localized Risk
Acronym: SHORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-A00042-51
Record Dates: First submitted 2017-12-07; First posted 2018-01-31 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: To Evaluate the Rate of Digestive and Urinary Toxicity
MeSH Terms: interventions — Brachytherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- brachytherapy + External radiotherapy (Experimental): Prostate booster, HDR brachytherapy with 15Gy in 1 fraction + external radiotherapy 25Gy in 5 fractions
  Interventions: Radiation: prostatic boost in brachytherapy with high dose rate (HDR)
- External radiotherapy (Active Comparator): Exclusive external radiotherapy. 25Gy in 5 fractions + a 40Gy prostate boost in stereotaxic conditions.
  Interventions: Radiation: prostatic boost in brachytherapy with high dose rate (HDR)

INTERVENTIONS:
Radiation: prostatic boost in brachytherapy with high dose rate (HDR) — prostatic boost in brachytherapy with high dose rate (HDR)

SUMMARY:
The standard treatment of high-risk prostatic adenocarcinoma is based on pelvic-prostatic external radiotherapy combined with concomitant and adjunctive hormone therapy for a total of 3 years.

Prostatic stereotactic radiotherapy in 5 sessions is a therapeutic option currently delivered and described in multiple cohorts of patients with a tolerance comparable to normo-fractional treatments. This therapeutic scheme makes it possible to deliver a higher equivalent biological dose than during a treatment carried out with a conventional fractionation.

The results with a follow-up of 9 years are extremely encouraging and do not show any excess toxicity compared to other irradiation techniques. They confirm that urinary and digestive toxicities are acceptable. All these studies did not involve pelvic irradiation. Several trials have also demonstrated the feasibility of normofractionated pelvic irradiation associated with hypofractionated prostatic irradiation using an integrated boost technique.

The primary objective is to evaluate, for localized high-risk prostate cancers (unfavorable intermediate or high risk), the rate of digestive and urinary toxicity cumulated at 3 months of the association of a pelvi-prostatic irradiation contracted in 5 sessions, with:To evaluate, for localized high-risk prostate cancers (unfavorable intermediate or high risk), the rate of digestive and urinary toxicity cumulated at 3 months of the association of a pelvi-prostatic irradiation contracted in 5 sessions, with:

* a prostatic boost in brachytherapy with high dose rate (HDR) or
* an integrated boost in stereotaxis (in case of contraindication to brachytherapy)

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the prostate
2. Patient with one of the following cases:

   * Gleason 7 - 10 + T1c - T2b + PSA < 50 ng/mL or
   * Gleason 6 + T2c - T4 ou envahissement ≥ 50% sur les biopsies + PSA < 50 ng/mL or
   * Gleason 6 + T1c - T2b + PSA > 20 ng/mL
3. Risk of lymph node involvement> 15%
4. Patient N0, or Nx
5. Prostate volume estimated on MRI or ultrasound less than 60 cc.
6. Absence of pelvic lymphadenopathy ≥ 15 mm on CT or MRI extension assessment
7. Lack of bone and / or visceral metastasis on CT scan and bone scintigraphy
8. Hormonal treatment started maximum 90 days before the beginning of the irradiation,
9. IPSS score <12 without alpha blocker treatment
10. Absence of prior pelvic radiotherapy,
11. Lack of surgical treatment for prostate cancer except transurethral resection performed within 6 months before radiotherapy,
12. Age ≥ 18 years and ≤ 85 years,
13. WHO performance index ≤ 1,
14. Estimated life expectancy> 5 years,
15. Indication of treatment with radiotherapy and validated hormone therapy in a multidisciplinary consultation meeting
16. Affiliation to a social security scheme,
17. Signed informed consent.

Exclusion Criteria:

1. Prostate cancer of histology other than adenocarcinoma,
2. Patient diagnosed with N1 during imaging or pN1,
3. serum PSA level> 100 ng / ml,
4. IPSS score ≥ 12 or alpha blocker treatment,
5. Prostate volume estimated on MRI or ultrasound> 60 cc
6. History of cancer in the 5 years prior to entry into the trial,
7. History of trans-urethral resection of prostate less than 6 months old,
8. History of rectal surgery,
9. History of pelvic irradiation,
10. Patient with severe hypertension not controlled by appropriate treatment,
11. Contraindication to pelvic irradiation,
12. Patient not eligible for brachytherapy

    * Prostate volume> 60cc
    * Urine flow measurement with max flow <12 mL / s
    * Or curative anticoagulant treatment
    * Or contraindication to general anesthesia
13. Patient treated with antineoplastic or drug may include methotrexate,
14. Hormone therapy started> 90 days before the first irradiation,
15. Patient on immunosuppressant therapy
16. Contraindication to agonists or antagonists of LHRH,
17. Bilateral hip prosthesis,
18. Patient already included in another therapeutic trial with an experimental molecule,
19. Patient unable to cooperate during treatment,
20. Persons deprived of their liberty or guardianship,
21. Inability to undergo medical follow-up of the test.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-24 (Actual); Primary Completion 2029-04-24 (Estimated); Study Completion 2029-04-24 (Estimated)

PRIMARY OUTCOMES:
The rate of digestive and urinary toxicity accumulated at 3 months | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Georges François Leclerc, Dijon
  - CGFL, Dijon